CLINICAL TRIAL: NCT05341336
Title: Outcome and Prognostic Factors of Surgical Management of Scalp Arteriovenous Malformations
Brief Title: Outcome and Prognostic Factors of Surgical Management of Scalp AVMs.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Antonios Bakheet Henis Soliman, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPFSMSAM
Record Dates: First submitted 2021-12-03; First posted 2022-04-22 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Cirsoid Aneurysm
MeSH Terms: conditions — Arteriovenous Malformations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical excision (Experimental): complete surgical excision of the scalp AVMs after identifying feeding arteries, vein and high flew shunts to perform a complete devascularization of the AVM.
  Interventions: Procedure: total surgical excision

INTERVENTIONS:
Procedure: total surgical excision — patients will be operated under general anesthesia. Pressure is applied along the incision line while staying away from the palpable margin of the AVM lesion and used Raney clips to control bleeding.
  Once the skin flap was raised, the lesion could be seen through the galea. The galea around the lesion is incised, and the lesion will be separated from the underlying skin using a combination of bipolar diathermy and sharp dissection.
  The nidus is often located in galeal aponeurosis. Dilated arteries and veins extended into subcutaneous tissue, which was separated with special care to prevent accidental nidus rupture and avoid excessive cauterization to prevent postoperative scalp necrosis.
  Ligation is applied on feeder arteries, then applied to veins with total excision of the lesion.
  After excision of the lesion, the skin flap was replaced with interrupted stitches.
  The wound was allowed to heal primarily along with intravenous administration of antibiotics.

SUMMARY:
Scalp arteriovenous malformations (AVMs) are rarely encountered vascular scalp anomalies that represent 8% of all AVMs. Different terms are being used to describe the vascular anomalies of the scalp include cirsoid aneurysm, racemosum aneurysm, plexiform angioma, arteriovenous fistula and arteriovenous malformation. Derived from the Greek language, kirsos, the term cirsoid aneurysm is used to describe the AVM as it resembles varix. Case studies reported approximately 200 cases with increased prevalence during the last 15 years. The etiology of scalp AVMs remains controversial, it can be spontaneous or traumatic. They generally develop in the trauma background and in patients over 30-year-old while spontaneous scalp AVM may present at birth and remains asymptomatic until adulthood.

DETAILED DESCRIPTION:
Patients with scalp AVMs are usually presented with scalp swelling, and cosmetic concerns along with other presentations including headache, pain, tinnitus, audible bruits, palpable thrills, and hemorrhage. Neuro-radiological diagnosis is the cornerstone for the surgical procedure to be performed, and cranial angiography is of great significance for diagnosis and treatment selection. MRA is also of significance for establishing a diagnosis as scalp AVMs are confused with hemangioma and cavernomas. Treatment of the cirsoid aneurysm is difficult due to the abnormal fistulous communications between the feeding arteries and veins and high shunt flow. Management protocols for scalp AVMs include various options including surgical excision, endovascular embolization, ligation, and intralesional injections. Operative blood loss, postoperative cosmetic complications are significant concerns when treating scalp AVMs, thus various methods are used pre and postoperatively in order to control these concerns. A thorough analysis of scalp AVMs regarding anatomy, feeder vessels, size, and other different variables is required for a better understanding of the problem in order to improve the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with scalp AVMs confirmed by various imaging techniques. AVMs of the scalp will include: cirsoid aneurysm, serpentinum aneurysm, racemosum aneurysm, plexiform angioma, arteriovenous fistula, high flow shunts and arteriovenous malformations.
* Age group: any age group.
* Aetiology: congenital, traumatic, or any.

Exclusion Criteria:

* High risk patients or unfit for surgery.
* Patients refused surgery, or scheduled for endovascular intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Occlusion of the feeding arteries and veins confirmation by imaging techniques | This will be monitored for a period of 6 months post-operative.
  identifying the occluded arteries and vein of the excised AVM through the use of diagnostic radiology including CT angiography and conventional angiography to evaluate the results of a well planned surgical excision of scalp AVM.
  This will be monitored for a period of 6 months post operative.
Cosmetic outcome according to the modified Hollandar scale | This will be monitored for a period of 6 months post-operative.
  Following up the cosmetic outcome according to the modified Hollandar scale to achieve better prognosis and higher patient satisfaction.
  The modified Hollandar scale: 0 score represents the best score, and an overall score of 6 points represents the worst outcome.
  the use of the modified Hollander scale would be used for post-operative evaluation and a period of 6 month-follow-up.

SECONDARY OUTCOMES:
Detect prognostic factors that affect the outcomes: etiology | This will be monitored for a period of 6 months post-operative.
  By identifying the important factors affecting the outcome including:
  etiology: congenital, traumatic or idiopathic. Studying how etiology can affect the outcome of surgical excision of scalp AVMs.
Detect prognostic factors that affect the outcomes: age | This will be monitored for a period of 6 months post-operative.
  By identifying the important factors affecting the outcome including:
  age Studying how age variation can affect the outcome of surgical excision of scalp AVMs and compare different age groups to prognosis.
Detect prognostic factors that affect the outcomes: site and size | This will be monitored for a period of 6 months post-operative.
  By identifying the important factors affecting the outcome including:
  site and size: the site and size of the scalp AVM and how the site affects the prognosis post-operative.
Detect prognostic factors that affect the outcomes: Primary arterial supply of the AVM, number of feeders | This will be monitored for a period of 6 months post-operative.
  By identifying the important factors affecting the outcome including:
  Primary arterial supply of the AVM, number of feeders: through the use of imaging techniques, determine the primary feeding arteries and their numbers and hw it will affect the prognosis and recurrence rate.
  Studying the distribution of the AVMs and their primary arterial supply and the number of feeding arteries and how this can affect the outcome of surgical excision of scalp AVMs.
  based on the anatomy of arterial supply.
Detect prognostic factors that affect the outcomes: clinical symptoms | This will be monitored for a period of 6 months post-operative.
  By identifying the important factors affecting the outcome including:
  clinical symptoms: how pre-operative symptoms could be indicative for prognosis compared to post-operative symptoms in case of any residuals.
  Studying various symptoms compared with post-operative residuals, if any, and how they can affect the outcome of surgical excision of scalp AVMs.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurkanlar D, Gonul M, Solmaz I, Gonul E. Cirsoid aneurysms of the scalp. Neurosurg Rev. 2006 Jul;29(3):208-12. doi: 10.1007/s10143-006-0023-y. Epub 2006 Apr 6. PMID 16598510
- [Background] Komiyama M, Nishikawa M, Kitano S, Sakamoto H, Imai K, Tsujiguchi K, Mizuno T. Non-traumatic arteriovenous fistulas of the scalp treated by a combination of embolization and surgical removal. Neurol Med Chir (Tokyo). 1996 Mar;36(3):162-5. doi: 10.2176/nmc.36.162. PMID 8869152
- [Background] Heilman CB, Kwan ES, Klucznik RP, Cohen AR. Elimination of a cirsoid aneurysm of the scalp by direct percutaneous embolization with thrombogenic coils. Case report. J Neurosurg. 1990 Aug;73(2):296-300. doi: 10.3171/jns.1990.73.2.0296. PMID 2366088
- [Background] Albuquerque Sousa LH, Maranha Gatto LA, Demartini Junior Z, Koppe GL. Scalp Cirsoid Aneurysm: An Updated Systematic Literature Review and an Illustrative Case Report. World Neurosurg. 2018 Nov;119:416-427. doi: 10.1016/j.wneu.2018.08.098. Epub 2018 Aug 24. PMID 30149169
- [Background] Sofela A, Osunronbi T, Hettige S. Scalp Cirsoid Aneurysms: Case Illustration and Systematic Review of Literature. Neurosurgery. 2020 Feb 1;86(2):E98-E107. doi: 10.1093/neuros/nyz303. PMID 31384940
- [Background] Furtado SV, Srinivasa R, Vala K, Mohan D. Contemporary management of scalp cirsoid aneurysm: A dual-trained neurosurgeon's perspective. Clin Neurol Neurosurg. 2021 Feb;201:106437. doi: 10.1016/j.clineuro.2020.106437. Epub 2020 Dec 15. PMID 33373833
- [Background] Li F, Zhu S, Liu Y, Chen Y, Chi L, Chen G, Zhang J, Qu F. Traumatic arteriovenous fistula of the superficial temporal artery. J Clin Neurosci. 2007 Jun;14(6):595-600. doi: 10.1016/j.jocn.2006.04.011. Epub 2007 Mar 26. PMID 17379525
- [Background] Mohamed WN, Abdullah NN, Muda AS. Scalp arteriovenous malformation : a case report. Malays J Med Sci. 2008 Jul;15(3):55-7. PMID 22570590
- [Background] Khodadad G. Arteriovenous malformations of the scalp. Ann Surg. 1973 Jan;177(1):79-85. doi: 10.1097/00000658-197301000-00015. No abstract available. PMID 4682507